CLINICAL TRIAL: NCT03498612
Title: Phase II Window Study of Pembrolizumab in Untreated B-Cell Non-Hodgkin Lymphoproliferative Diseases
Brief Title: Pembrolizumab in Untreated B-Cell Non-Hodgkin Lymphoproliferative Diseases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed per SRC Low Accrual Policy.
Sponsor: University of Washington (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ajay Gopal, Professor, Division of Medical Oncology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9647; NCI-2018-00432 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9647 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1716072 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-03-27; First posted 2018-04-13 (Actual); Results first posted 2022-12-30 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Follicular Lymphoma; Indolent B-Cell Non-Hodgkin Lymphoma; Marginal Zone Lymphoma
Keywords: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 18 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with B-cell non-Hodgkin lymphoproliferative diseases that have not been treated. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 18 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Must have measurable disease defined by at least one of the following criteria:

  * Lesions greater than 1.5 cm that can be accurately measured in two dimensions by computed tomography (CT) (preferred), or magnetic resonance imaging (MRI)
* Must have indication for treatment (adapted from National Comprehensive Cancer Network [NCCN] 2015 guidelines)

  * Any of the following constitute an indication for treatment:
  * Significant symptoms due to any iBCL: Which may include pain/discomfort, limitation of function, fatigue/malaise/constitutional symptoms, B-symptoms (fever, weight loss, night sweats), pruritus
  * Threatened end-organ function due to any iBCL
  * Progressive cytopenia secondary to any iBCL
  * Steady progression of follicular lymphoma (FL) and marginal zone lymphoma (MZL)
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 500/uL Note: Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed. No lower limit if cytopenia is related to bone marrow involvement.
* Platelets >= 25000/uL Note: Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed. No lower limit if cytopenia is related to bone marrow involvement.
* Hemoglobin >= 8 g/dL Note: Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed. No lower limit if cytopenia is related to bone marrow involvement.
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN (GFR can also be used in place of creatinine or CrCl)

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN ( =< 5 x ULN for participants with liver metastases)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had prior chemotherapy, radiation therapy, or immunotherapy for the diagnosis of iBCL
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Be in urgent need of therapy for lymphoma related complications (such as hyperviscosity syndrome) and those with bulky disease
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K. Gopal, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (pembrolizumab): Patients receive pembrolizumab 200mg IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 18 cycles in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
Period: Overall Study
Arm/Group | Treatment (pembrolizumab)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 55 [39 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete Response [CR] + Partial Response [PR] for Follicular Lymphoma and Marginal Zone Lymphoma)
Description: Measured by Lugano Criteria evaluated by positron emission tomography (PET)/computed tomography (CT) or CT or white blood cell count for chronic lymphocytic leukemia (CLL). The corresponding 95% two-sided confidence interval will be derived.
Time Frame: Up to 8 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (pembrolizumab)
Number analyzed (Participants) | 9
Participants | 3

2. Secondary Outcome: Duration of Response
Description: Kaplan Meier methodology will be used to estimate event-free curves.
Time Frame: From the time by which the measurement criteria are met for CR or PR, whichever is recorded first, until death or the first date by which recurrent or progressive disease is objectively documented, assessed up to 5 years
Measure: Mean (Full Range); unit: Months
Arm/Group | Treatment (pembrolizumab)
Number analyzed (Participants) | 9
Months | 41 [4 to 60]

3. Secondary Outcome: Progression-free Survival
Description: Data for subjects without disease progression or death will be censored at the date of the last tumor assessment. Kaplan-Meier methodology will be used to estimate the event-free curves.
Time Frame: From the first study drug administration to the first occurrence of lymphoma progression or death from any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (pembrolizumab)
Number analyzed (Participants) | 9
Months | 6.3 [3.77 to NA] — The upper limit of the 95% confidence interval could not be estimated due to insufficient number of participants with events.

4. Secondary Outcome: Time to Next Therapy
Time Frame: From the time of first study drug administration until the date of the first subsequent therapy given to treat the indolent B-cell non-Hodgkin lymphoproliferative diseases, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (pembrolizumab)
Number analyzed (Participants) | 9
Months | 5.4 [4.73 to NA] — The upper limit of the 95% confidence interval could not be estimated due to insufficient number of participants with events.

5. Secondary Outcome: Count of Participants Who Experience Adverse Events (AEs)
Description: Safety summaries will include tabulations in the form of tables. The frequency of treatment-emergent AE's will be summarized. Additional AE summaries will include AE frequency by AE severity and relationship to the study drug.
Time Frame: Up to 90 days after last dose, up to 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (pembrolizumab)
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: From the time of informed consent through 90 days following the last dose of pembrolizumab, up to 1 year.
Description: Method of routinely determining whether or not certain adverse events have occurred happen through regular investigator assessment, regular laboratory testing, and patient self-reporting.
Arm/Group | Treatment (pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (pembrolizumab) (N=9)
Rituximab Desensitization Protocol (General disorders) | 1 (1)
Retroperitoneal Venous Hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (pembrolizumab) (N=9)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
ACTH decreased (Endocrine disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (6)
Alkaline phosphatase increased (Investigations) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dry Eye (Eye disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Elevated TSH (Endocrine disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Fever (General disorders) | 1 (1)
Elevated T3 (Endocrine disorders) | 1 (1)
Elevated T4 (Endocrine disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (4)
Left shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Right forehead pink papule (Skin and subcutaneous tissue disorders) | 1 (1)
Right lower rib pain (General disorders) | 1 (1)
Scrotal edema (Reproductive system and breast disorders) | 1 (1)
Left foot fungal infection (Infections and infestations) | 1 (1)
Testosterone decreased (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT03498612/Prot_SAP_000.pdf